CLINICAL TRIAL: NCT01800331
Title: Text2bHealthy: Enhancing Adherence to Childhood Obesity Treatment Through the Use of Innovative Methods
Brief Title: Text2bHealthy: Using Innovative Methods in Childhood Obesity Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: My post-doctoral fellow did not return from her mat leave and I have no other students to take on this project.
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-03175
Record Dates: First submitted 2013-02-18; First posted 2013-02-27 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text2bHealthy (Experimental): The intervention arm receives the Text2bHealthy program on a PDA
  Interventions: Behavioral: Text2bHealthy
- Control group (No Intervention): The control group will complete a paper dairy to keep track of their lifestyle behaviours

INTERVENTIONS:
Behavioral: Text2bHealthy — The intervention group uses handheld computers to keep track of their lifestyle behaviours and they will receive feedback on thier progress and tips (Text2bHealthy)
  Arms: Text2bHealthy

SUMMARY:
In Canada, the number of obese children and adolescents has increased tremendously. Interventions addressing diet and physical activity have been successful in the short-term. However, a great number of individuals have difficulties maintaining achieved weight loss and returning to treatment sessions.

New technology interventions, through the web or delivered trough Personal Digital Assistants (PDAs) (e.g. iPhone or Blackberry), are increasingly being used in health interventions. PDAs have emerged as appealing in health interventions as they are easily accessible and their interactivity makes them well suited to promote long-term engagement in behaviour change interventions.

This study will look at the utility of supplementing a family-based lifestyle program for overweight and obese adolescents (Shapedown BC) with a PDA intervention (Text2bHealthy) focussing mainly on physical activity, sedentary behaviours, and dietary intake to maintain treatment success by improving self-management skills. Adolescents and will receive Text2bHealthy for 3-months after 3 months participation in the Shapedown BC program.

Results from this study will provide needed information on how to improve treatment adherence and maintenance outcomes through the use of innovative methods and will ultimately contribute to the improvement of long-term outcomes in obesity treatment.

DETAILED DESCRIPTION:
Around the world, the amount of people who are overweight is increasing. This has become a public health crisis. Obesity, especially in children, is a problem because it is associated with risk for health problems and psychological issues. These problems include heart disease and poor quality of life and can happen both in childhood and later life.

Programs that help people change their lifestyle and behaviour are effective to help people lose weight and improve their mental health. In children, the main issue for treating obesity is to help the child keep weight off and to prevent a return to unhealthy behaviours. This means that long-term support is needed. But the health care system is not set up to do this because of a limited amount of resources. The aim of this study is to see if there are better long-term results if we use a technology tool along with a lifestyle program.

The aim of this study is to examine a personal digital assistant (PDA) program (Text2bHealthy) supplemented to an existing family-based group treatment for overweight and obese children. This treatment is called the British Columbia Centre for Healthy Weights (BCCHW) Shapedown BC program. The aim of this study is to see if Text2bHealthy supplemented to the Shapedown BC program helps children to keep the weight of and improves physical activity as well as fruit, vegetable, and fat intake.

We know from studies that reporting one's own behaviour, goal setting, and tailored feedback are key elements in changing health behaviours. Text2bHealthy includes these key elements. PDAs will be given to 30 10-16 year old children and adolescents after completing the Shapedown BC program. They will be explained how to use the PDA. Children who participate in the Text2bHealthy program will set weekly goals related to their physical activity, eating or sitting behaviours. Also, they will report on their lifestyle behaviours twice a week. They will receive personalized feedback on their progress. The feedback is designed to be supportive and to reinforce their behaviour in a positive way. The control group (N=30) will use a paper dairy to keep track of their lifestyle behaviours. At 0 and 3 months after completing the Shapedown BC program, measurements such as height and weight will be taken. Also, exercise and nutrition behaviour will be measured. Physical activity will be measured with pedometers and a recall and nutrition intake with questionnaires.

Because it is hard to maintain weight loss, we need to provide programs that offer the long-term support of behaviour change. Tools such as PDAs seem to be ideal to offer long-term support. For the purpose of this study, PDAs will be used as a proof of concept; the programming can be incorporated into smart phones in the future. From previous studies we know that reporting one's own behaviour seems to improve weight loss in children. Also, behaviours are more likely to be reported when using mobile phones compared to paper & pencil diaries. I am one of the first to study the effect of innovative technologies by using self-reporting, goal setting, and personalized feedback in childhood obesity treatment. We hope that the results from this study will increase our knowledge on the use and feasibility of digital devices in childhood obesity treatment.

The outcomes of this research will be used to better understand how to improve weight loss maintenance among obese children. Obesity places children at higher risk for heart disease and poor quality of life when they are adults. Thus time and cost-effective long-term support programs need to be developed to improve weight loss maintenance. This new program has the potential to improve maintenance of weight loss and healthy lifestyle in overweight and obese children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese teens
* Aged 10 to 16 years
* Completion of the Shapedown BC program
* Being a resident of the greater metropolitan area of Vancouver
* Not expected to move within the study time period
* Ability to read and speak in English at a 6th grade level

Exclusion Criteria:

* Participating in other physical activity or nutrition studies or programs such as the Weight Watchers or Jenny Craig
* Pregnancy
* Any co-morbidities which require immediate medical attention
* Any musculoskeletal, cardiovascular, pulmonary, or orthopedic problems or disabilities precluding from being physically active
* Use of a prescription medication which could interfere with the child's weight
* Failure to complete the Shapedown BC program
* Diagnosis of Type 1 diabetes

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
BMI-z scores | 3 months

SECONDARY OUTCOMES:
Physical activity (physical activity recall, questions and pedometer steps) | 3 months
Nutrition | 3 months
Sitting behaviour (recall) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Louise Masse, PhD, Principal Investigator — University of British Columbia
Locations (1):
- The British Columbia Children's Hospital, Vancouver, British Columbia, Canada